CLINICAL TRIAL: NCT02911987
Title: Structural and Functional Effects of High Intensity Training (HIT) Program in Patients With Non-specific Chronic Low Back Pain. A Randomized Clinical Trial
Brief Title: Structural and Functional Effects of High Intensity Training (HIT) Program in Patients With Non-specific Chronic Low Back Pain
Acronym: LBP-HIT-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Annick Timmermans, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LBP-HIT-RCT
Record Dates: First submitted 2016-09-13; First posted 2016-09-23 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- the 'cardio' HIT group (Experimental): Group 1 receives HIT exercise, aimed only at improving cardiovascular endurance (the 'cardio' HIT group).
  Interventions: Other: high intensity training (HIT) program
- the 'general' HIT group (Experimental): Group 2 receives HIT exercise aimed at improving both cardiovascular and general muscle condition (the 'general' HIT group ).
  Interventions: Other: high intensity training (HIT) program
- the 'lumbar' HIT group (Experimental): Group 3 receives HIT exercise, aimed at improving both cardiovascular condition and specific trunk muscle condition (the 'lumbar' HIT group).
  Interventions: Other: high intensity training (HIT) program
- the 'combined' HIT group (Experimental): Group 4 receives HIT exercise which is a combination of previous programs (cardiovascular fitness, muscular fitness and general training specific trunk muscles) (the 'combined' HIT group). These trainings will take place in the REVAL Rehabilitation Research Center on the campus of Hasselt University in Diepenbeek.
  Interventions: Other: high intensity training (HIT) program
- control group (Active Comparator): Group 5 receives MIT exercise consisting of a combination of previous programs (cardiovascular fitness, muscular fitness and general training specific trunk muscles) (the 'MIT' group)
  Interventions: Other: moderate intensity training (MIT) exercise therapy

INTERVENTIONS:
Other: high intensity training (HIT) program — The participants are randomly divided through use of sealed envelopes into four groups that all follow high intensity training (HIT) programs. Each training group follows of a 12 week program (2x/week, 2h). All training will be conducted under the guidance of expert therapists.
  Arms: the 'cardio' HIT group; the 'combined' HIT group; the 'general' HIT group; the 'lumbar' HIT group
Other: moderate intensity training (MIT) exercise therapy — MIT exercise consisting of a combination of previous programs (cardiovascular fitness, muscular fitness and general training specific trunk muscles) (the 'MIT' group).
  Arms: control group

SUMMARY:
Low back pain is a common disorder, occurring worldwide in both males and females in all age groups. The prevalence is higher in females and the incidence peaks between 30 and 65 years. It is currently the most frequent musculoskeletal cause of functional disability and it has a major socio-economic impact on today's society. Although a small percentage of persons with low back pain can be diagnosed with a specific underlying cause, almost 90% of persons with low back pain present with symptoms of nonspecific origin. A part of these symptoms are only of short duration, but 23% of all people will develop nonspecific chronic low back pain (NSCLBP).

Exercise therapy (ET) is currently an important component in the treatment of NSCLBP. Previous studies analysed the effects of various modes of exercise therapy, such as motor control therapy, core stability training and aerobic conditioning training. However, therapy outcomes can be low, and guidelines in favour of using a specific program are contradictory. It thus still remains unclear which therapy modality is best suited. Furthermore, no recommendations are available about optimal training intensities during rehabilitation of persons with NSCLBP.

Since as well aerobic as muscular deconditioning are apparent in persons with chronic low back pain and improvements in overall physical fitness can affect therapy outcomes in this population, ET specifically focussing on physical fitness can be advocated for NSCLBP rehabilitation. High Intensity Training (HIT), has been promoted as an effective and efficient training method for improving physical fitness and health related parameters in healthy persons. Also, HIT resulted in successful reconditioning and improvement of functional and disease related outcomes in persons with other chronic diseases such as multiple sclerosis, heart failure, COPD and cardiometabolic diseases. Although some studies showed promising results for the effect of HIT on low back pain such as high intensity isolated, evidence is still scarce and study results are unclear because of methodological shortcomings.

The aim of this randomized clinical trial study is to evaluate the effects of a HIT program on disease related outcomes, physical fitness and muscle contractile characteristics compared to a conventional rehabilitation program in persons with NSCLBP.

ELIGIBILITY:
Inclusion Criteria:

1. medically diagnosed with non-specific chronic low back pain,
2. over 25 years old,
3. Oswestry Disability Index: disability score >20%,
4. able to understand Dutch (spoken and written),
5. Physical Activities Scale For Individuals with Physical Disabilities <30. -

Exclusion Criteria:

1. invasive surgery at the lumbar spine in the last 18 months (arthrodesis was excluded, microsurgery was allowed),
2. radiculopathy (uni- or bilateral),
3. co-morbidities: paresis and/or sensory disturbances by neurological causes, diabetes mellitus, rheumatoid arthritis, an increase of pain of 3 points with a result of > 8/10 on the Numeric Pain Rating Scale (NPRS) in the last 48 hours, pregnancy,
4. ongoing compensation claims and/or (work)disability > 6 months,
5. rehabilitation/exercise therapy program for LBP in the past 6 months. -

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
pain | day 1
  The Numeric Pain Rating Scale (NPRS) is a nominal scale on which the participant indicates the amount of pain he/she perceives at that current moment. It consists of a line indicating eleven successive scores (0-10), whereby score 0 means 'no pain' and score 10 means 'worst pain imaginable'. An improvement of 2 levels or more is accepted as clinically relevant.
pain | week 6
  The Numeric Pain Rating Scale (NPRS)
pain | week 12
  The Numeric Pain Rating Scale (NPRS)
Kinesiophobia | day 1
  The Tampa Scale for Kinesiophobia (TSK) is an ordinal 17 item questionnaire that inventories pain-related fear of movement for persons with subacute and chronic low back pain or fibromyalgia. A higher score relates to more pain-related fear.
Kinesiophobia | week 6
  The Tampa Scale for Kinesiophobia (TSK) is an ordinal 17 item questionnaire that inventories pain-related fear of movement for persons with subacute and chronic low back pain or fibromyalgia. A higher score relates to more pain-related fear.
Kinesiophobia | week 12
  The Tampa Scale for Kinesiophobia (TSK) is an ordinal 17 item questionnaire that inventories pain-related fear of movement for persons with subacute and chronic low back pain or fibromyalgia. A higher score relates to more pain-related fear.
Physical disability RMDQ | day 1
  The Roland Morris Disability Questionnaire (RMDQ) is an ordinal 24 item questionnaire for evaluating the disability level of the patient with low back pain with regards to activities of daily living. A higher score correlates to a higher level of disability and a change of 5 is the minimal clinically important difference.
Physical disability RMDQ | week 6
  The Roland Morris Disability Questionnaire (RMDQ) is an ordinal 24 item questionnaire for evaluating the disability level of the patient with low back pain with regards to activities of daily living. A higher score correlates to a higher level of disability and a change of 5 is the minimal clinically important difference.
Physical disability RMDQ | week 12
  The Roland Morris Disability Questionnaire (RMDQ) is an ordinal 24 item questionnaire for evaluating the disability level of the patient with low back pain with regards to activities of daily living. A higher score correlates to a higher level of disability and a change of 5 is the minimal clinically important difference.
Endurance capacity | day 1
  Endurance capacity is tested to volitional fatigue on an electronically braked bike ergometer
Endurance capacity | week 6
  Endurance capacity is tested to volitional fatigue on an electronically braked bike ergometer
Endurance capacity | week 12
  Endurance capacity is tested to volitional fatigue on an electronically braked bike ergometer
Abdominal/back strength | day 1
  The maximum voluntary isometric and dynamic strength of back and abdominal muscles is measured using an isokinetic dynamometer (System 3, Biodex, Enraf-Nonius, New York).
Abdominal/back strength | week 6
  The maximum voluntary isometric and dynamic strength of back and abdominal muscles is measured using an isokinetic dynamometer (System 3, Biodex, Enraf-Nonius, New York).
Abdominal/back strength | week 12
  The maximum voluntary isometric and dynamic strength of back and abdominal muscles is measured using an isokinetic dynamometer (System 3, Biodex, Enraf-Nonius, New York).
Muscle Biopsy | day 1
  muscle biopsies of the paravertebral muscles of the spine are obtained through a micro biopsy procedure (Biopsy gun, Bard Medical). This is done by a trained physician with extensive experience in taking muscle biopsies. The obtained muscle samples are divided into cryovials, per subject and per measurement (for the determination of muscle fiber CSA, muscle fiber characterization, distribution, angiogenesis, muscle fiber characteristics, etc.).
  Safety Issue: Yes, taking a piece of muscle tissue, can be slightly painful, but there are no serious risks involved. There will be no permanent damage to the muscle. The risk of infection in the wound can never be excluded. However, the site of the biopsy is thoroughly decontaminated and sealed in order to achieve a good wound healing and prevent an infection. A local bleeding may occur in the muscle causing a bruise.
Muscle Biopsy | week 12
  muscle biopsies of the paravertebral muscles of the spine are obtained through a micro biopsy procedure (Biopsy gun, Bard Medical). This is done by a trained physician with extensive experience in taking muscle biopsies. The obtained muscle samples are divided into cryovials, per subject and per measurement (for the determination of muscle fiber CSA, muscle fiber characterization, distribution, angiogenesis, muscle fiber characteristics, etc.).
  Safety Issue: Yes, taking a piece of muscle tissue, can be slightly painful, but there are no serious risks involved. There will be no permanent damage to the muscle. The risk of infection in the wound can never be excluded. However, the site of the biopsy is thoroughly decontaminated and sealed in order to achieve a good wound healing and prevent an infection. A local bleeding may occur in the muscle causing a bruise.
Physical disability ODI | day 1
  The Modified Oswestry Disability Index (ODI) is a valid and reliable questionnaire for evaluating constraints experienced by people in their daily activities due to chronic low back pain. It consists of 10 items that are scored on a 5-point scale. The total score gives a percentage degree of limitation for the patient.
Physical disability ODI | week 6
  The Modified Oswestry Disability Index (ODI) is a valid and reliable questionnaire for evaluating constraints experienced by people in their daily activities due to chronic low back pain. It consists of 10 items that are scored on a 5-point scale. The total score gives a percentage degree of limitation for the patient.
Physical disability ODI | week 12
  The Modified Oswestry Disability Index (ODI) is a valid and reliable questionnaire for evaluating constraints experienced by people in their daily activities due to chronic low back pain. It consists of 10 items that are scored on a 5-point scale. The total score gives a percentage degree of limitation for the patient.
activity level | day 1
  Physical Activities Scale For Individuals with Physical Disabilities (PASIPD) The PASIPD is a questionnaire consisting of 13 items to measure the physical activity of people with disabilities. It provides information about leisure, household and work-related physical activity in the last 7 days.
activity level | week 6
  Physical Activities Scale For Individuals with Physical Disabilities (PASIPD) The PASIPD is a questionnaire consisting of 13 items to measure the physical activity of people with disabilities. It provides information about leisure, household and work-related physical activity in the last 7 days.
activity level | week 12
  Physical Activities Scale For Individuals with Physical Disabilities (PASIPD) The PASIPD is a questionnaire consisting of 13 items to measure the physical activity of people with disabilities. It provides information about leisure, household and work-related physical activity in the last 7 days.

SECONDARY OUTCOMES:
Body composition | day 1
  The body composition is obtained by means of a dual Energy X-Ray Absorptiometry (DEXA) scan.
Body composition | week 6
  The body composition is obtained by means of a dual Energy X-Ray Absorptiometry (DEXA) scan.
Body composition | week 12
  The body composition is obtained by means of a dual Energy X-Ray Absorptiometry (DEXA) scan.
physical activity tracking | day 1
  Activity of the daily routine will be evaluated by means of wearing an accelerometer (Actigraph GT3X activity monitors) (2 midweek days and 1 weekend day, 3 consecutive days) throughout the day. A schedule will be inventoried by the participant (diary).
physical activity tracking | week 12
  Activity of the daily routine will be evaluated by means of wearing an accelerometer (Actigraph GT3X activity monitors) (2 midweek days and 1 weekend day, 3 consecutive days) throughout the day. A schedule will be inventoried by the participant (diary).
disability in participation and quality of life | day 1
  Short Form Health Survey (SF-36) The SF-36 is a 36 item scale that assesses eight health concepts (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health) with the possibility of independent scoring for each.
disability in participation and quality of life | week 6
  Short Form Health Survey (SF-36) The SF-36 is a 36 item scale that assesses eight health concepts (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health) with the possibility of independent scoring for each.
disability in participation and quality of life | week 12
  Short Form Health Survey (SF-36) The SF-36 is a 36 item scale that assesses eight health concepts (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health) with the possibility of independent scoring for each.
Motivation VAS | day 1
  The start motivation is measured by a visual analog scale (VAS).
Motivation IMI | day 1
  At the end of the study setting viewing detailed motivation for the program based on the Intrinsic Motivation Inventory (IMI) (on T1).
Motivation VAS | week 6
  The start motivation is measured by a visual analog scale (VAS).
Motivation IMI | week 6
  At the end of the study setting viewing detailed motivation for the program based on the Intrinsic Motivation Inventory (IMI) (on T1).
Motivation VAS | week 12
  The start motivation is measured by a visual analog scale (VAS).
Motivation IMI | week 12
  At the end of the study setting viewing detailed motivation for the program based on the Intrinsic Motivation Inventory (IMI) (on T1).

CONTACTS AND LOCATIONS:
Overall Officials: Annick Timmermans, prof. dr., Principal Investigator — Hasselt University; Frank Vandenabeele, prof. dr., Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided